CLINICAL TRIAL: NCT04358900
Title: Unobtrusive Monitoring of Affective Symptoms and Cognition Using Keyboard Dynamics
Brief Title: Unobtrusive Monitoring of Affective Symptoms and Cognition Using Keyboard Dynamics (UnMASCK)
Acronym: UnMASCK
Status: Active, not recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Olusola Alade Ajilore, Principal Investigator, University of Illinois at Chicago
Other Study IDs: 2019-1333; 1R01MH120168-01A1 (NIH)
Record Dates: First submitted 2020-04-08; First posted 2020-04-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Mood Disorders; Major Depressive Disorder; Bipolar Disorder I; Bipolar Disorder II; Persistent Depressive Disorder (Dysthymia); Cyclothymia
MeSH Terms: conditions — Mood Disorders; Depressive Disorder, Major; Bipolar Disorder; Dysthymic Disorder; Cyclothymic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mood disorder group: Participants must meet criteria for one of the following disorders according to Diagnostic and Statistical Manual of Mental Disorders-5 criteria (52): major depressive disorder (MDD), persistent depressive disorder (PDD), bipolar disorder (BD) type I/type II, cyclothymia. Multiple mood disorders are employed, in line with the Research Domain Criteria (RDoC; (53)) framework and the relative imprecision of current symptom diagnostic clusters for tracking treatment responses and course of disease. To ensure adequate representation across diagnostic categories (including controls), the investigators will cap enrollment of major mood disorders (MDD, BD type I/II) to 50%, PDD and cyclothymia to 25% and recruit a healthy comparison group to comprise the remaining 25% of the sample.
- Control group: Participants who do not meet the Diagnostic and Statistical Manual of Mental Disorders-5 criteria for (52): major depressive disorder (MDD), persistent depressive disorder (PDD), bipolar disorder (BD) type I/type II, or cyclothymia.

SUMMARY:
Mood disorders are associated with significant financial and health costs for the United States, partially due to cognitive problems in these patients that can worsen disease course and impair treatment response. This study proposes to use smartphone-based technology to monitor cognitive problems in patients with mood disorders by linking brain network changes with predicted worsening of mood symptoms. The proposed study will provide evidence for using smartphone-based passive sensing as a cost-effective way to predict illness course and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* 25-50 years, as age-related declines in brain connectivity occur starting around 40-45 years of age (49-51);
* Participants must meet criteria for one of the following disorders according to Diagnostic and Statistical Manual of Mental Disorders-5 criteria (52): major depressive disorder (MDD), persistent depressive disorder (PDD), bipolar disorder (BD) type I/type II, cyclothymia. To ensure adequate representation across diagnostic categories (including controls), the investigators will cap enrollment of major mood disorders (MDD, BD type I/II) to 50%, PDD and cyclothymia to 25% and recruit a healthy comparison group to comprise the remaining 25% of the sample.
* Own a BiAffect-compatible smartphone.

Exclusion Criteria:

* Active suicidal ideation as determined by the Columbia Suicide Severity Rating Scale (C-SSRS)(50), suicide attempt in the last 3 months
* Severe cognitive impairment secondary to a neurological disorder (mild cognitive impairment, neurocognitive disorders, traumatic brain injury, developmental delay)
* Active moderate or severe alcohol and/or substance use disorders;
* Major medical or neurologic illness that would interfere with protocol adherence and/or interpretation of findings; and
* Presence of contraindications to MRI.
* Pregnancy (positive pregnancy test), trying to become pregnant, or lactation.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will recruit 132 participants (100 with mood disorders, and 32 controls) from the Chicago area, psychiatry clinics at the UIC, and longitudinal studies of Dr. Langenecker (MH091811 and MH 101487). All subjects will be recruited using community outreach efforts, not limited to but including listserv emails, flyers, word of mouth, and health fairs.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging | Change from week 2 to week 4.
  a. Neuroimaging based biomarkers of cognitive performance will include Structural brain network Efficiency Interhemispheric Efficiency, Reduced nodal efficiency in ventrolateral prefrontal cortex/altered modularity, Reduced nodal efficiency in anterior cingulate cortex, and Reduced nodal efficiency in salience networks. Neuroimaging will take place while the participant completes the parametric Go/No-go test completed during a functional magnetic resonance imaging after using BiAffect app for 2 weeks, and again after using the BiAffect app for 4 weeks.
BiAffect Metric | Measured at the end of week 4 after using the BiAffect app for 4 weeks
  1. BiAffect Metric component 1, Typing speed: Data collected through the keyboard provided by the BiAffect app to measure the Average Interkey Delay (The average time between keystrokes measured in seconds) and keys per second will be combined to report typing speed.
  2. BiAffect Metric component 2, Backspace Ratio: Data collected through the keyboard provided by the BiAffect app to measure the number of backspace keypresses divided by total keypresses.
  3. BiAffect Metric component 3, Autocorrect Rate: Data collected through the keyboard provided by the BiAffect app to measure the number of autocorrect events divided by total keypresses. These 3 components will be combined to report the BiAffect Metric.
Clinical symptoms | Measured at baseline.
  1. Severity of depressive symptoms: In person administration of the Inventory of Depressive Symptomatology (IDS-C/QIDS-C). Possible scores range from 0-111 where higher scores indicate more severe depression symptoms.
  2. Symptoms of mania: In person administration of the Young Mania Rating Scale (YMRS) which has a total score range from 0 to 60; higher scores indicate a more severe mania.
  3. Symptoms of depression: In person administration of the Hamilton Rating Scale for Depression (HAM-D). Scores range between 0-52, and the higher the score the more depressive symptoms a participant has. These questionnaires will be combined to produce the clinical symptoms measure.
Cognition | Change from week 2 to week 4
  1. Attention/ processing speed will be measured in person using the Flanker Inhibitory Control and Attention Test (scores range 0-5, and higher scores mean better attention), the Pattern Comparison Processing Speed Test (scores range 0-130, and higher scores mean faster processing speed), and the Trail Making Task part A (scores range 0-300 seconds, and lower scores mean faster processing speed).
  2. Cognitive control will be measured in person using the Dimensional Change Card Sort Test (scores range 0-10, and higher scores mean better cognitive control), the Flanker Inhibitory Control and Attention Test, and the Trail Making Task part B (scores range 0-300 seconds, and lower scores mean higher cognitive control).
  3. Working memory will be measured in person using the List Sorting Working Memory Test (scores range 0-28, and higher scores mean better working memory). Attention, cognitive control, and working memory scores will be combined to produce the cognitive outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Olusola Ajilore, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No